CLINICAL TRIAL: NCT00574379
Title: A Multi-Center Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Once or Twice Daily Bilastine (10 or 20 mg) Compared With Placebo Given Orally in The Treatment of the Symptoms of Seasonal Allergic Rhino-Conjunctivitis With Allergy to Mountain Cedar Pollen
Brief Title: Efficacy, Safety and PK of Once or Twice Daily Bilastine (10 or 20 mg) Compared With Placebo in the Symptomatic Treatment of SAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Allied Research International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA 2607/RAE; CTFZ07001
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Seasonal Allergic Rhinitis; Hay Fever; Allergic Conjunctivitis; Hypersensitivity
Keywords: Allergic Rhinitis; Mountain Cedar Pollen; Pollen Allergy; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic; Hypersensitivity; Rhinitis, Allergic | interventions — bilastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Bilastine 20mg once per day
  Interventions: Drug: Bilastine
- 2 (Experimental): Bilastine 20mg twice per day
  Interventions: Drug: Bilastine
- 3 (Experimental): Bilastine 10mg once per day
  Interventions: Drug: Bilastine
- 4 (Experimental): Bilastine 10mg twice per day
  Interventions: Drug: Bilastine
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — Bilastine 10 or 20mg, once or twice daily for 14 days. Tablets
  Arms: 1; 2; 3; 4
Drug: Placebo — Placebo tablets twice daily for 14 days
  Arms: 5

SUMMARY:
Evaluate the relative efficacy of four dosing regimens of bilastine tablets (given either once or twice per day) versus placebo in patients with Seasonal Allergic Rhinitis (SAR) in the Mountain Cedar season in south Texas and Oklahoma based on the mean change from baseline in Reflective Total Nasal Symptom Scores (TNSS) assessed over 14 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical history of Seasonal Allergic Rhinoconjunctivitis with seasonal onset and offset of nasal allergy symptoms
* documentation of a positive skin test within one year of screening to Mountain Cedar allergen

Exclusion Criteria:

* significant medical condition
* significant nasal abnormality
* significant cardiac condition
* recent infection
* use of other allergy medication during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in nasal symptom scores | 14 days

SECONDARY OUTCOMES:
Change in ocular symptom scores and quality of life scores; standard safety assessments | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ander Sologuren, MD, Study Director — Faes Farma, S.A.; Paul Ratner, MD, Principal Investigator — Sylvana Research Associates
Locations (13):
- United States (13):
  - Oklahoma Allergy and Asthma Clinic, Oklahoma City, Oklahoma
  - MetaClin Research Inc., Austin, Texas
  - Austin Clinical Research, Austin, Texas
  - Lovelace Scientific Resources, Austin, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - DGD Research, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Southwest Allergy and Asthma Centre, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Live Oak Allergy and Asthma, San Antonio, Texas
  - Allergy & Asthma Care of Waco, Waco, Texas
  - Allergy Asthma Research Institute, Waco, Texas